CLINICAL TRIAL: NCT02228434
Title: Study on the Tailored Intervention Strategy of Childhood Obesity Based on Monitoring Physical Activities and Dietary Behaviors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wang Jingjing (Other)
Responsible Party: Sponsor-Investigator, Wang Jingjing, Institute of Child and Adolescent Health, Peking University
Organization: Peking University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB00001052-10081
Record Dates: First submitted 2014-08-27; First posted 2014-08-29 (Estimated); Last update posted 2014-08-29 (Estimated); Status verified 2014-08

CONDITIONS: Pediatric Obesity
Keywords: Childhood obesity, intervention, effectiveness, comparison
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (4):
- Tailored intervention group (Experimental): For the monitoring session, physical activity was assessed by accelerometer and dietary was assessed by diary. Based on the monitoring information, the individual tailored prescription, including the normative feedback and process feedback, were formed and delivered to children and parents. Children were encouraged to modify the behaviors according to the prescription.
  Then, next monitoring circle was followed. In total, 7 monitoring round were completed.
  Interventions: Behavioral: Monitoring and Tailored prescription; Behavioral: General Health Education
- Happy 10 exercise group (Experimental): All the schools participating in this group were encouraged to take two Happy 10 sessions on each school day.
  Interventions: Behavioral: Happy 10 program; Behavioral: General Health Education
- Nutrition education group (Experimental): The nutrition intervention was mainly conducted based on the nutrition knowledge through health education lectures given by researchers. The lectures were given for eight times to students and twice to parents. Each lecture session lasted no less than 40 min.
  Interventions: Behavioral: Specified nutrition education; Behavioral: General Health Education
- Control group (No Intervention): Receive no intervention

INTERVENTIONS:
Behavioral: Monitoring and Tailored prescription
  Other Names: ZhiJi accelerometer UX-02 as physical activity monitor
  Arms: Tailored intervention group
Behavioral: Happy 10 program
  Other Names: happy 10 program developed by Center for Disease Control and Prevention, China
  Arms: Happy 10 exercise group
Behavioral: Specified nutrition education
  Arms: Nutrition education group
Behavioral: General Health Education
  Arms: Happy 10 exercise group; Nutrition education group; Tailored intervention group

SUMMARY:
The project aims at developing the tailored intervention strategy of childhood obesity based on monitoring physical activities with accelerometer and dietary behaviors using diary. It probably raise the passion of obese children to control weight, form healthy life style, be effective in sustaining weight loss and early prevent adulthood diseases.

DETAILED DESCRIPTION:
The overweight and obese primary school students from 1-5 grades will be recruited according to "Body Mass Index Reference for Screening Overweight and Obesity in Chinese School-age Children". The participants with will be allocated with schools as the unit to four groups: tailored intervention based on monitoring physical activity and dietary behaviors, exercise intervention group based on the Happy 10 program, nutrition education intervention group. The three intervention groups received the designed interventions for the duration of 1 year. Before and after the intervention, we will carry out a questionnaire survey, a physical measurement, a fitness test, and a metabolic markers detection

ELIGIBILITY:
Inclusion Criteria:

* Overweight and obese children from grade 1-5 primary schools

Exclusion Criteria:

* Students with any contraindication or physical diseases (heart, Lung, liver, kidney, other vital organs, endocrine diseases and drug side effects et al.) and psychological illnesses that may prevent them from participating in physical activity and eating a normal diet were excluded

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 450 (Actual)
Dates: Start 2009-05; Primary Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Change in body mass index | Baseline, 1-year post-intervention

SECONDARY OUTCOMES:
Change in obesity-related anthropometric measurements | Baseline, 1-year post-intervention
Change of blood pressure | Baseline, 1-year post-intervention
Change of biomarkers for disease risk | Baseline, 1-year post-intervention
Change of attitude, knowledge, and behaviors on dietary and physical activity | Baseline, 1-year post-intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Insitute of Child and Adolescent Health, Peking University, Beijing, China

REFERENCES:
- [Derived] Wang JJ, Lau WC, Wang HJ, Ma J. Evaluation of a comprehensive intervention with a behavioural modification strategy for childhood obesity prevention: a nonrandomized cluster controlled trial. BMC Public Health. 2015 Dec 3;15:1206. doi: 10.1186/s12889-015-2535-2. PMID 26635229